CLINICAL TRIAL: NCT01377909
Title: An Investigator-initiated Pilot Study Using Statins to Improve the Anti-HCV Response to Peginterferon Alfa 2-b and Ribavirin in Previous Non-responders
Brief Title: HCV Treatment With Fluvastatin, Simvastatin to Improve Interferon Sensitivity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator retiring
Sponsor: Bader, Ted, M.D. (Individual)
Responsible Party: Principal Investigator, Ted Bader, MD, Director of Liver Diseases, Professor, Department of Medicine, Section of Gastroenterology, Bader, Ted, M.D.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Bader 15859
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C, interferon
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- statin (Experimental)
  Interventions: Drug: statin

INTERVENTIONS:
Drug: statin — daily statin orally for 48 weeks

SUMMARY:
Objective: The goal is to improve peginterferon sensitivity in previous poor responders. "Sensitivity" here means the host's ability to kill more HCV.

Design: Twenty poor responders to prior PIFN/RBV will be given 48 weeks of statin monotherapy. Veterans and civilians between the ages of 18 and 70 are eligible.

ELIGIBILITY:
Inclusion Criteria:

Hepatitis C positive by HCV RNA within 180 days. - No anti-HCV medicine within 30 days of screening

Exclusion Criteria:

* decompensated liver disease
* severe cardiac disease (ejection fraction < 20% or uncontrolled angina)
* unexplained muscle pain at time of screening
* pregnancy
* renal insufficiency (creatine clearance < 50 ml/min)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Improvement in peginterferon response as measured by change in HCV RNA levels | 48 weeks
  The change in hepatitis C viral load in response to one injection of peginterferon will be measured with a baseline pre-study viral load and response to an injection of peginterferon; this test will be remeasured 48 weeks later. The change in viral loads over time will be assessed statistically.

SECONDARY OUTCOMES:
The response of interferon stimulated genes | 48 weeks
  The number of known interferon activated genes will be assessed by microarray from serum samples at baseline and then reassessed by microarray 48 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Ted Bader, M.D., Principal Investigator — VA Medical Center
Locations (1):
- Veterans Administration Medical Center (VAMC), Oklahoma City, Oklahoma, United States